CLINICAL TRIAL: NCT04174612
Title: A Phase 3, Prospective, Randomized Multi-center Intervention Trial of Early Intensification in AML Patients Bearing FLT3 Mutations Based on Peripheral Blast Clearance: A MYNERVA-GIMEMA Study
Brief Title: AML Patients Bearing FLT3 Mutations Based on Peripheral Blast Clearance
Acronym: AMELIORATE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML1919
Record Dates: First submitted 2019-11-11; First posted 2019-11-22 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation
MeSH Terms: interventions — Cytarabine; Daunorubicin; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard clinical treatment (Active Comparator): Patients will complete "3+7" + Midostaurin induction course.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Midostaurin
- Experimental treatment (Experimental): The experimental arm will provide 2 main modifications compared to standard:
  i) immediate switch to intensified induction with high-doses Cytarabine (on days 5, 6 and 7 of induction) ii) early allocation to high-risk disease category to be refined according to ELN stratification and post induction MRD status
  Interventions: Drug: Daunorubicin; Drug: Midostaurin; Drug: Cytarabine HD

INTERVENTIONS:
Drug: Cytarabine — 100 mg/m2/bid day 1-3 100 mg/m2/die day 4-7
  Arms: Standard clinical treatment
Drug: Daunorubicin — 60 mg/m2/die day 1-3
Drug: Midostaurin — 50 mg/bid day 8-21
Drug: Cytarabine HD — 100 mg/m2/bid day 1-3 100 mg/m2/die day 4 1.500 mg bid day 5-7
  Arms: Experimental treatment

SUMMARY:
Prospective, multi-center, interventional, randomized, open clinical trial for the treatment of acute myeloid leukemia with FLT3 mutations customized upon the prognostic parameter PBC

ELIGIBILITY:
Inclusion Criteria:

1. Patients with de novo AML, untreated, newly diagnosed, according to WHO 2016 criteria
2. Presence of a mutation of FLT3 gene, either ITD and/or TKD
3. Adequate availability of diagnostic biologic material for full cytological, cytogenetic, genetic and immunophenotypic disease characterization according to ELN criteria.
4. Presence of morphologically identifiable blasts on peripheral blood at diagnosis
5. Presence of a Leukemia-associated aberrant immune-phenotype (LAIP) as assessed by MFC (multiparametric flow cytometry) at diagnosis
6. Age between 18 and 65 years, included
7. ECOG performance status 0-2 or disease-related reversible ECOG 3 score following adequate supportive care.
8. Signed written informed consent according to ICH/EU/GCP and national local laws

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia
2. Diagnosis of AML with t(8;21)(q22:q22)/RUNX1-RUNX1T1 and t(16;16)(p13:q22) or inversion of chromosome 16 (16)(p13q22)/CBFB-MYH11; in case of suspicion of CBF-related AML due to morphological and/or immunophenotypic features, specific FISH or molecular testing is strongly recommended in accordance with WHO criteria3,157
3. Patients with LVEF less than 45% (by echocardiogram or MUGA)
4. Pre-existing, uncontrolled pathology such as heart failure (congestive/ischaemic, acute myocardial infarction within the post 3 months, untreatable arrhythmias, NYHA classes III and IV), sever liver disease with total bilirubin ≥2,5 x ULN and/or ALT>3 ULN (unless attributable to AML), acute or chronic pancreatitis, kidney function impairment with serum creatinine ≥2,5 (unless attributable to AML) and severe neuropsychiatric disorder that impairs the patient's ability to understand and sign the informed consent or to cope with the intended treatment plan. For altered liver, pancreas and kidney function tests, eligibility criteria can be reassessed at 24-96 hours, following the institution of adequate supportive measures.
5. Uncontrolled bacterial or fungal infections
6. QTc >470 msec on screening ECG (Fridericia's formula)
7. A history of cancer that is not in remission phase following surgery and/or chemotherapy and/or radiotherapy with life expectancy < 1 year.
8. Pregnancy declared by the patient herself. A pregnancy test is performed at diagnosis and, if applicable, before allogeneic HSCT . Female and male patients who are fertile must agree to use an effective form of contraception with their sexual partners from enrollment through 4 months after the end of treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 2,5 years
  Improvement of outcome measured as event-free survival (EFS) in patients with FLT3+ acute myeloid leukemia who are predicted to have low chemosensitivity, as defined upon the biomarker "peripheral blast clearance (PBC)", following the application of an early intensification of overall treatment, both in induction (high-doses delivery) and in consolidation (allocation to allogeneic transplant) phase, compared with standard regimens

SECONDARY OUTCOMES:
Adverse events rate | 2,5 years
  Adverse events rate according to CTCAE criteria
Rate of death in aplasia | 2 months
  rate of death in aplasia
Neutrophil recovery | 2 months
  Median number of days for neutrophil recovery
platelet recovery | 2 months
  Median number of days for platelet recovery
CR rate | 6 months
  Complete remission rate after induction
DFS | 2 years
  Disease-free survival
OS | 2 years
  Overall survival
CIR | 2 years
  Cumulative incidence of relapse
MRD assessment | 6 months
  MRD negativity rate at the end of induction and consolidation

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (20):
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Irccs Oncologico Istituto Tumori Giovanni Paolo Ii - Bari - Uo Ematologia, Bari
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Aou Careggi- Sod Ematologia, Florence
  - Asl Latina, Presidio Ospedaliero Nord - Ospedale Santa Maria Goretti - Uoc Ematologia, Latina
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Aou San Luigi Gonzaga - Orbassano - Scdu Ematologia Generale E Oncoematologia, Orbassano
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - Aou Policlinico P. Giaccone - Palermo - Uo Ematologia, Palermo
  - Fondazione Ircss Policlinico San Matteo - Pavia - Uo Ematologia, Pavia
  - Ausl Della Romagna, Ospedale "Santa Maria Delle Croci" - Ravenna - Ematologia, Ravenna
  - Grande Ospedale Metropolitano "Bianchi-Melacrino-Morelli" Po E. Morelli - Reggio Calabria - Uoc Ematologia, Reggio Calabria
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - C.R.O.B. - I.R.C.C.S. - Rionero in Volture - Uoc Ematologia, Rionero in Vulture
  - Aou Policlinico Tor Vergata - Roma - Uoc Trapianto Cellule Staminali, Roma
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Ospedale Mauriziano Umberto I - Torino - Scdu Ematologia, Torino